CLINICAL TRIAL: NCT06079164
Title: A Phase 1 Open-label, Single Arm, Multicenter Study Evaluating the Safety and Efficacy of KITE-197 in Subjects With Relapsed or Refractory Large B-cell Lymphoma
Brief Title: Study of KITE-197 in Participants With Relapsed or Refractory Large B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-656-0601
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Large B-cell Lymphoma
MeSH Terms: conditions — Recurrence | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KITE-197 (Experimental): Phase 1a (Dose Escalation): Participants with r/r large B-cell lymphoma will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by a single target starting dose of KITE-197 chimeric antigen receptor (CAR) transduced autologous T cells. Based on dose limiting toxicities (DLTs) observed in the first cohort, additional participants will be enrolled and administered escalating dose of KITE-197.
  Phase 1b (Dose Expansion): After completion of dose escalation, additional participants with r/r B-cell lymphoma across different disease indications will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine followed by a single dose of KITE-197 CAR-transduced autologous T cells at 1 or more dose-level deemed to be tolerable.
  Interventions: Drug: KITE-197; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: KITE-197 — A single infusion of CAR-transduced autologous T cells administered intravenously
Drug: Cyclophosphamide — Lymphodepleting chemotherapy administered intravenously
Drug: Fludarabine — Lymphodepleting chemotherapy administered intravenously

SUMMARY:
This study will have two Phases: Phase 1a and Phase 1b. The goal of Phase 1a of this clinical study is to learn more about the safety, tolerability and dosing of study drug KITE-197, in participants with relapsed or refractory large B-cell lymphoma (r/rLBCL). The goal of Phase 1b of this clinical study is learn about the effectiveness of the recommended dose of KITE-197 in participants with r/r LBCL.

The primary objectives of this study are:

Phase 1a: To evaluate the safety of KITE-197 in participants with r/r LBCL and determine the target dose level for Phase 1b.

Phase 1b: To evaluate the efficacy of KITE-197 in participants with r/r LBCL as measured by the complete remission (CR) rate.

DETAILED DESCRIPTION:
Participants will be followed for approximately 6 months after the infusion of KITE-197 before transitioning to a separate Kite long-term follow-up study KT-US-982-5968, in which they will be followed for the remainder of the 15-year follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

* Relapsed or Refractory Large B-cell Lymphoma
* At least 1 measurable lesion
* Adequate organ and bone marrow function

Key Exclusion Criteria:

* History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (eg, cervix, bladder, breast) unless disease free for at least 2 years
* History of Richter's transformation of chronic leukemic lymphoma
* History of allogenic stem cell transplant (SCT)
* Autologous SCT within 6 weeks of planned KITE-197 infusion
* Prior CD19 targeted antibody, such as tafasitamab and loncastuximab with the exception of individuals who have previously achieved an objective response to such therapy and their tumor expresses CD19 by International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (IHC) at the time of screening. Individuals who meet these criteria may be eligible
* Prior treatment with bendamustine within 6 months of enrollment
* Prior CAR therapy or other genetically modified cell therapy
* Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management
* History of HIV infection or acute or chronic active hepatitis B or C infection
* History or presence of a clinically significant central nervous system (CNS) disorder Note: Prior or active CNS involvement by lymphoma is not an exclusion criterion.
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, New York Heart Association Class II or greater congestive heart failure, or other clinically significant cardiac disease within 12 months before enrollment
* Presence of primary immunodeficiency
* History of autoimmune disease (eg, Crohn's disease, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years
* History of symptomatic deep vein thrombosis (DVT) or pulmonary embolism within 3 months before enrollment. Catheter induced DVT which has been treated for at least 6 weeks prior to enrollment is permitted
* Females of childbearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Percentage of Participants Experiencing any Dose-limiting Toxicities (DLTs) | First infusion date of KITE-197 up to 28 days
Phase 1b: Complete Remission (CR) Rate | Up to 24 months
  Complete remission rate is defined as the proportion of participants with complete remission, per international working group (IWG) Lugano classification, as assessed by the investigator.

SECONDARY OUTCOMES:
Percentage of Participants Experiencing Adverse Events (AEs) | Enrollment up to 24 months plus 30 days
Percentage of Participants Experiencing Serious Adverse Events (SAEs) | Enrollment up to 24 months plus 30 days
Overall Response Rate (ORR) | Up to 24 months
  ORR is defined as the proportion of participants with best objective response of either a CR or a partial response (PR) during the trial prior to any new anti-lymphoma therapy, per the Lugano Classification, as determined by the investigator.
Duration of Response (DOR) | Up to 24 months
  DOR is defined as the time from first objective response to disease progression or death from any cause among participants who have achieved CR or PR per the Lugano Classification, as determined by the investigator.
Progression-Free Survival (PFS) | Up to 24 months
  PFS is defined as the time from KITE-197 infusion to disease progression per the Lugano Classification, as determined by investigator review or death from any cause.
Event Free Survival (EFS) | Up to 24 months
  EFS is defined as the time from KITE-197 infusion to the earliest occurrence of death due to any cause, disease progression/relapse per investigator, or initiation of new anti-lymphoma therapy.
Time to Next Treatment (TTNT) | Up to 24 months
  TTNT is defined as time from KITE-197 infusion to the start of subsequent new lymphoma therapy or death from any cause.
Overall Survival (OS) | Up to 24 months
  OS is defined as the time from KITE-197 infusion to death from any cause.
Number of KITE-197 CAR T Cells in Blood Over Time Post Infusion | Up to 24 months
Proportion of Immune Cell Subsets in KITE-197 | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (11):
- United States (5):
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Brisbane and Women's Hospital, South Brisbane, Queensland
  - The Alfred Hospital, Melbourne, Victoria
- Canada (3):
  - Cross Cancer Institute, Edmonton
  - QEII Health Sciences Centre, Halifax
  - Jewish General Hospital, Montreal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06079164